#### The GlaxoSmithKline group of companies

| Division | | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for Study 201499: A randomised, placebo-controlled, double-blind, two period crossover study to characterise the exhaled nitric oxide time profile as a biomarker of airway inflammation in adult asthma patients following repeat administration of inhaled Fluticasone Furoate (FF)/ Vilanterol (VI) 100/25 mcg |
|---|---|---|
| <b>Compound Number</b> | : | GW685698+GW642444 |
| Effective Date | : | 11-Apr-2017 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2015N241692 00
- The planned analyses and output to be included in Clinical Pharmacology Study Report for Protocol 201499. This RAP is intended to describe the pharmacodynamic, biomarker, safety and tolerability analyses required for the study which will be provided to the study team members to convey the content of the reporting efforts, specifically Statistical Analysis Complete (SAC).

#### **Author's Name and Functional Area:**

| PPD | | 31-Mar-2017 |
|-----------------|---------------|-------------|
| Associate Stati | stician (QSI) | 31-Wai-2017 |

#### Approved by:

| PPD | | 11 4 2017 |
|--------------|--------|-------------|
| Manager, Sta | istics | 11-Apr-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | | | PAGE NO. |
|---|---|---|---|---|
| 1. | REPC | RTING & | ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SLIMI | MARY OF I | KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | | pjective(s) and Endpoint(s) | |
| | 2.2. | | | |
| | | | esign | |
| | 2.4. | Statistica | al Hypotheses | |
| 3. | PLAN | NED ANA | LYSES | 8 |
| | 3.1. | Interim A | nalyses | 8 |
| | 3.2. | Final Ana | alyses | 8 |
| 4. | ΔΝΔΙ | YSIS POP | PULATIONS | q |
| •• | 4.1. | | Deviations | |
| | 7.1. | 1 1010001 | Deviations | |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | 40 |
| | CON | ENTIONS | S | 10 |
| 6. | STUD | Y POPUL | ATION ANALYSES | 11 |
| ٥. | 6.1. | | v of Planned Analyses | |
| | 0.1. | OVCIVICV | Voi i lailitea Allaiyses | |
| 7. | PRIM | ARY STAT | FISTICAL ANALYSES | 12 |
| | 7.1. | Pharmac | codynamic Analyses | 12 |
| | | 7.1.1. | Overview of Planned Pharmacodynamic Analyses | |
| | | | 7.1.1.1. Statistical Analysis of Pharmacodynamic | |
| | | | Parameters | |
| | | 7.1.2. | Planned Primary Pharmacodynamic Statistical Analyses | s13 |
| 8. | SECC | NDARY S | STATISTICAL ANALYSES | 13 |
| - | 8.1. | | codynamic Analyses | |
| | <b>0</b> | 8.1.1. | Overview of Planned Pharmacodynamic Analyses | |
| | | 8.1.2. | Planned Secondary Pharmacodynamic Statistical Analyses | |
| | | 0.1.2. | Trainied Secondary Tharmacodynamic Statistical Analyses | |
| 9. | | R STATIS | STICAL ANALYSES | 15 |
| | 9.1. | | v of Planned Biomarker Analyses | |
| | | 9.1.1. | Overview of Planned Analyses | 15 |
| | 9.2. | Overview | v of Safety Analyses | 16 |
| | | 9.2.1. | Overview of Planned Adverse Events Analyses | 16 |
| | | 9.2.2. | Overview of Planned Clinical Laboratory Analyses | |
| | | 9.2.3. | Overview of Planned Other Safety Analyses | |
| 10. | REFE | RENCES. | | 18 |
| 11 | APPE | NDICES | | 10 |
| | 11.1. | | x 1: Protocol Deviation Management and Definitions for F | |
| | | | Population | |
| | 11.2. | Appendix | x 2: Data Management | 21 |
| | 11.3. | Appendix | x 3: Time & Events | 22 |
| | | | x 4: Treatment States and Phases | |

#### CONFIDENTIAL

| 20 | ۱1 | 4 | a | ( |
|----|----|---|---|---|

| | 11.4.1. | Treatment States for AE Data | 25 |
|---|---|---|---|
| 11.5. | Appendix | c 5: Data Display Standards & Handling Conventions | 26 |
| | 11.5.1. | Study Treatment & Sub-group Display Descriptors | 26 |
| | 11.5.2. | Baseline Definition & Derivations | |
| | | 11.5.2.1. Baseline Definitions | 26 |
| | | 11.5.2.2. Derivations and Handling of Missing Baseline | |
| | | Data | 26 |
| | 11.5.3. | Reporting Process & Standards | 27 |
| 11.6. | Appendix | c 6: Derived and Transformed Data | 29 |
| | 11.6.1. | General | |
| | 11.6.2. | Study Population | 29 |
| | 11.6.3. | Pharmacodynamic | 30 |
| 11.7. | Appendix | 7: Premature Withdrawals & Handling of Missing Data | 31 |
| | 11.7.1. | Premature Withdrawals | 31 |
| | 11.7.2. | Handling of Missing Data | 31 |
| | | 11.7.2.1. Handling of Missing Dates | 31 |
| | | 11.7.2.2. Handling of Partial Dates | 32 |
| | | 11.7.2.3. Handling of Missing Data for Statistical | |
| | | Analysis | 32 |
| 11.8. | Appendix | 8: Model Checking and Diagnostics for Statistical | |
| | Analyses | | 33 |
| | | Statistical Analysis Assumptions | |
| 11.9. | | (9 – Abbreviations & Trade Marks | |
| | 11.9.1. | Abbreviations | |
| | 11.9.2. | Trademarks | |
| 11.10. | | 10: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverable [Priority] | |
| | | Study Population Tables | |
| | | Pharmacodynamic Tables | |
| | | Pharmacodynamic Figures | |
| | | Safety Tables | |
| | | Biomarker Tables | |
| | | Biomarker Figures | |
| | | .ICH Listings | |
| | | Non-ICH Listings | |
| 11.11. | Appendix | c 11: Example Mock Shells for Data Displays | 44 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol GlaxoSmithKline Document Number 2015N241692_00 |
| | • The planned analyses and output to be included in Clinical Pharmacology Study Report for Protocol 201499. This RAP is intended to describe the pharmacodynamic, biomarker, safety and tolerability analyses required for the study which will be provided to the study team members to convey the content of the reporting efforts, specifically Statistical Analysis Complete (SAC). |
| Protocol | • Reporting and Analysis Plan is based on original protocol (Dated: [12-JAN-2016]) for study 201499 [GlaxoSmithKline Document Number: 2015N241692_00] |
| Primary<br>Objective /<br>Endpoint | To characterise the fraction of exhaled nitric oxide (FeNO) time profile following repeat administration of fluticasone furoate/vilanterol (FF/VI) 100/25mcg combination in comparison with placebo in subjects with asthma as measured by: Change from baseline FeNO over time following the cessation of repeat dose treatment with FF/VI. |
| Secondary<br>Objective/<br>Endpoint | Change in FeNO over the treatment period following repeat administration of FF/VI 100/25mcg combination in comparison with placebo in subjects with asthma measured by: |
| | Change from baseline FeNO over the FF/VI treatment period. |
| | To determine the Peak Expiratory Flow (PEF) during and following repeat administration of FF/VI 100/25mcg combination in comparison with placebo in subjects with asthma measured by: |
| | Measurement of PEF during treatment and following cessation of repeat dose treatment with FF/VI. |
| | To determine forced expiratory volume in 1 second (FEV1) following repeat administration of FF/VI 100/25mcg combination in comparison with placebo in subjects with asthma as measured by: |
| | • Measurement of FEV1 pre-treatment and for up to 7 days after cessation of repeat dose treatment with FF/VI. |

| Overview | Key Elements of the RAP |
|---|---|
| Exploratory<br>Objective /<br>Endpoint | To investigate the effect of repeat administration of FF/VI 100/25mcg combination on exploratory biomarkers, including but not limited to, blood eosinophil levels and serum periostin levels, in comparison with placebo in subjects with asthma as measured by: |
| | Measurement of exploratory biomarkers, including but not limited to, blood eosinophil and serum periostin levels at baseline, and at various time points after cessation of repeat dose treatment with FF/VI |
| Study<br>Design | Randomised, double blind, placebo-controlled, two-period, crossover repeat dose study in adult subjects with asthma. |
| | Approximately twenty eight adult asthmatic subjects will be enrolled to ensure 24 subjects complete dosing and critical assessments for both treatment periods. |
| | Each subject will participate in two treatment periods of 14 (+ 2 days). FF/VI 100/25mcg will be received once daily (AM dosing) in one period and placebo (AM dosing) will be administered in the other period. At the end of each treatment period, there will be a monitoring period of 21 days. Following the 21 day monitoring period following treatment period 1, there may be a period of up to a further 4 weeks before the subjects start treatment period 2. |
| Planned<br>Analyses | <ul> <li>No interim analysis is planned.</li> <li>The final planned analyses will be performed after database freeze has been declared.</li> </ul> |
| Analysis<br>Population | <ul> <li>All Subjects Population comprise of all subjects randomised to treatment who received at least one dose of study medication</li> <li>Pharmacodynamic Population comprise of all Subjects in the 'All Subjects' population who had at least one PD assessment</li> </ul> |
| Hypothesis | No formal hypothesis will be tested, an estimation approach will be adopted to address the primary objective. A point estimate and corresponding 95% CI will be constructed for the treatment ratio of test treatment, $\mu(\text{test})$ and reference treatment, $\mu(\text{reference})$ , where FF/VI $100/25\text{mcg}$ is the test treatment and placebo the reference treatment |
| Primary<br>Analyses | FeNO, change from baseline ratio will be formally analysed following loge-transformation. A mixed effects repeated measures model will be fitted with fixed effect terms for period, treatment, day, time, (period-level baseline)*day*time interaction term, treatment*day*time interaction term, period-level baseline and subject-level baseline. Day*time interaction term will be fitted as repeated measure. FeNO will be loge-transformed prior to deriving subject-level baseline and period-level baseline. |

| Overview | Key Elements of the RAP |
|---|---|
| Secondary<br>Analyses | FeNO change from baseline ratio during treatment and FEV1 will be analysed similarly to the primary FeNO endpoint. FEV1 will not be log- |
| Anaryses | transformed prior to analysis. |
| | PEF will be summarised. |
| Safety | Safety data will be summarized |
| Analyses | |
| Biomarker<br>Analyses | Exploratory endpoints of biomarkers will be summarized |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol [Dated: 12-JAN-2016].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary (Pharmacodynamic) | Primary (Pharmacodynamic) |
| To characterise the fraction of exhaled nitric oxide (FeNO) time profile following repeat administration of fluticasone furoate/vilanterol (FF/VI) 100/25mcg combination in comparison with placebo in subjects with asthma. | Change from baseline FeNO over time following the cessation of repeat dose treatment with FF/VI. |
| Secondary (Pharmacodynamic) | Secondary (Pharmacodynamic) |
| Change in FeNO over the treatment period following repeat administration of FF/VI 100/25mcg combination in comparison with placebo in subjects with asthma. | Change from baseline FeNO over the FF/VI treatment period |
| To determine the Peak Expiratory Flow (PEF) during and following repeat administration of FF/VI 100/25mcg combination in comparison with placebo in subjects with asthma. | Measurement of PEF during treatment and following cessation of repeat dose treatment with FF/VI. |
| To determine FEV1 following repeat administration of FF/VI 100/25mcg combination in comparison with placebo in subjects with asthma | Measurement of FEV1 pre-treatment and for up to 7 days after cessation of repeat dose treatment with FF/VI |

| Objectives | Endpoints |
|---|---|
| Exploratory (Biomarker) | Exploratory (Biomarker) |
| To investigate the effect of repeat | Measurement of exploratory biomarkers, |
| administration of FF/VI 100/25mcg | including but not limited to, blood |
| combination on exploratory biomarkers, | eosinophil and serum periostin levels at |
| including but not limited to, blood | baseline, and at various time points after |
| eosinophil levels and serum periostin levels, | cessation of repeat dose treatment with |
| in comparison with placebo in subjects with | FF/VI |
| asthma | |

## 2.3. Study Design



| Overview of Study Design and Key Features | |
|---|---|
| Treatment | Subjects will be randomized to one of two sequences AB or BA. |
| Assignment | Where, A=Placebo and B=FF/VI 100/25mcg. |
| | Subjects will be administered the first treatment in the sequence in the first |
| | period and the second treatment in the sequence in the second period. |

# 2.4. Statistical Hypotheses

No formal hypothesis will be tested, an estimation approach will be adopted to address the primary objective. A point estimate and corresponding 95% CI will be constructed for the treatment ratio of test treatment,  $\mu$  (test) and reference treatment,  $\mu$  (reference), where, FF/VI 100/25mcg is the test treatment and placebo the reference treatment.

#### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No interim analysis is planned.

# 3.2. Final Analyses

| Analysis | Details |
|---|---|
| Final Analyses | The final planned analyses will be performed after all subjects have completed the study and after database freeze/unblinding. See Section 6 Section 9 for all final planned analyses for this study. |

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release has been declared by Data Management.
- 3. All protocol deviations have been confirmed
- 4. All criteria for unblinding the randomisation codes have been met.
- 5. Randomisation codes have been distributed according to RandAll NG procedures.
- 6. Database freeze has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses/Endpoint(s)<br>Evaluated |
|---|---|---|
| Screened Subjects | Comprise of all subjects who attended the screening visit | Study Population |
| All Subjects<br>Population | Comprise of all subjects randomised to treatment who received at least one dose of study medication. | <ul><li>Study Population</li><li>Biomarker</li><li>Safety</li></ul> |
| Pharmacodynamic Population | Subjects in the 'All Subjects' population who had at least one PD assessment | <ul><li>Pharmacodynamic</li><li>FeNO</li><li>FEV1</li><li>PEF</li></ul> |

**NOTES:** Please refer to Appendix 10which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed by the study team prior to database release to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - o The SI dataset will include all protocol deviations, the analysis dataset will include only important protocol deviations. The analysis dataset will be used for the listing and summary of important protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided.
- The study endpoints will be reported using the populations detailed in Section 4 of this document regardless of whether the subjects deviate from the protocol.
- If there are subjects with protocol deviations that may potentially impact the PD endpoints which needs to be confirmed prior to unblinding, exploratory sensitivity analyses may be considered. It further sensitivity analyses of the data are produced, they will be detailed in the clinical study report.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Data Management |
| 11.3 | Appendix 3: Time and Event |
| 11.4 | Appendix 4: Treatment States and Phases |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 11.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| 11.9 | Appendix 9: Abbreviations & Trade Marks |
| 11.10 | Appendix 10: List of Data Displays |
| 11.11 | Appendix 11: Example Mock Shells for Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Endpoint | Data I | Data Displays Generated | |
|---|---|---|---|
| | Table | Figure | Listing |
| <b>Subject Disposition</b> | | | |
| Subject Disposition for the Subject Conclusion Record | Y | | |
| Reasons for Subject Withdrawal | | | Y |
| Screening Status and Reasons for Screen Failure | Y | | Y |
| Subjects Enrolled by Country and Site ID | Y | | |
| Subjects for Whom the Treatment Blind was Broken | | | Y |
| Planned and Actual Treatments | | | Y |
| <b>Protocol Deviations</b> | | | |
| Important Protocol Deviations | Y | | Y |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Y |
| Populations Analysed | | | |
| Study Populations | Y | | |
| Subjects Excluded from Any Population | | | Y |
| <b>Demographic and Baseline Characteristics</b> | | | |
| Demographic Characteristics | $Y^{[1]}$ | | Y |
| Age Ranges | Y | | |
| Race and Racial Combinations | Y | | $Y^{[2]}$ |
| <b>Prior and Concomitant Medications</b> | | | |
| Current & Past Medical Conditions | | | Y |
| Concomitant Medications | | | Y |
| Exposure | | | |
| Exposure to Study Treatment | Y | | Y |

#### **NOTES:**

- Y = Yes display generated.
- [1] Conditional Display for PD Population.
- [2] Listing of race.

### 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Pharmacodynamic Analyses

Statistical Analysis of Pharmacodynamic endpoints will be performed by or under the direct auspices of, Clinical Statistics, GlaxoSmithKline.

### 7.1.1. Overview of Planned Pharmacodynamic Analyses

The primary Pharmacodynamic analyses will be based on the "Pharmacodynamic (PD)" population, unless otherwise specified.

Table 3 provides an overview of the planned Pharmacodynamic analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 3 Overview of Planned Pharmacodynamic Analyses

| Endpoint | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sumr | nary | Individual | | Summary | | Individual | |
| | T | F | F | L | T | F | F | L |
| FeNo | Y | | | Y | Y | | | |

| Endpoint | Log <sub>e</sub> transformed | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Sta | ats Analy | ysis Summary | | | Individual | | |
| | T | F | L | T | F | L | F | L |
| FeNO | Y | Y | Y | Y | | | Y | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TF related to any summaries (descriptive statistics) of the observed raw data. Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.1.1. Statistical Analysis of Pharmacodynamic Parameters

For the PD parameter of FeNO, the following summary statistics will be calculated and tabulated by treatment:

- Untransformed Data: N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum, maximum
- **Log**<sub>e</sub>-transformed Data: Geometric mean, 95% CI for the geometric mean, SD of log<sub>e</sub>-transformed data and %CVb

### 7.1.2. Planned Primary Pharmacodynamic Statistical Analyses

#### **Primary Statistical Analyses**

#### **Endpoint**

• Change from baseline ratio of log<sub>e</sub> transformed FeNO over time following the cessation of repeat dose treatment with FF/VI.

#### **Model Specification**

Endpoints will be statistically analysed using a mixed models repeated measures (MMRM) model.

Terms fitted in the MMRM model will include:

Fixed effect terms: Period, Treatment, Day, Time, Period-level baseline\*Day\*Time interaction term, Treatment\*Day\*Time interaction term, Period-level baseline and Subject-level baseline.

Repeated: Day\*Time interaction term.

**Note**: FeNO will be log<sub>e</sub>-transformed prior to deriving subject-level baseline and period-level baseline.

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics will be performed for mentioned Statistical Analyses as required.

#### **Model Results Presentation**

- Point estimates and their associated 95% confidence intervals will be constructed for the difference [FF/VI 100/25mcg] – [Placebo] at each timepoint (AM and PM i.e. pre-dose & 12 hours) on each day. The point estimates and their associated 95% confidence intervals will then be back-transformed to provide point estimates and 95% confidence intervals for the ratios, [FF/VI 100/25mcg]/[Placebo] for each day and AM/PM timepoint.
- Estimates of within-subject variability for FeNO will also be provided, where  $CVw(\%) = SQRT(exp(MSE) 1) \times 100$  and MSE is the residual mean squared error from the model. CVw represents a pooled measure of within-subject variability across the regimens FF/VI 100/25mcg, Placebo and timepoints.

## 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Pharmacodynamic Analyses

#### 8.1.1. Overview of Planned Pharmacodynamic Analyses

The secondary Pharmacodynamic analyses will be based on the "Pharmacodynamic (PD)" population, unless otherwise specified.

Table 4 provides an overview of the planned Pharmacodynamic analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 4 Overview of Planned Pharmacodynamic Analyses

| Endpoint | Absolute | | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Summary Individual | | Stats Analysis | | | Summary | | Individual | | | |
| | T | F | F | L | T | F | L | T | F | F | L |
| FeNO <sup>[1]</sup> | | | | | Y | Y | Y | | | | |
| FEV1 | Y | | | Y | Y | Y | Y | Y | | | |
| PEF | Y | | | Y | | | | | | | |

#### **NOTES:**

[1] FeNO will be loge transformed prior to analysis.

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TF related to any summaries (descriptive statistics) of the observed raw data.

Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.1.2. Planned Secondary Pharmacodynamic Statistical Analyses

#### **Secondary Statistical Analyses**

#### **Endpoint**

• Change from baseline ratio of loge transformed FeNO during treatment with FF/VI.

#### **Model Specification**

Endpoints will be statistically analysed using a mixed models repeated measures (MMRM) model.

Terms fitted in the MMRM model will include:

Fixed effect terms: Period, Treatment, Day, Time, Period-level baseline\*Day\*Time interaction term, Treatment\*Day\*Time interaction term, Period-level baseline and Subject-level baseline.

Repeated: Day\*Time interaction term.

**Note**: FeNO will be log<sub>e</sub>-transformed prior to deriving subject-level baseline and period-level baseline.

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics will be performed for mentioned Statistical Analyses as required.

#### **Model Results Presentation**

- Point estimates and their associated 95% confidence intervals will be constructed for the difference [FF/VI 100/25mcg] [Placebo] at each timepoint (AM/PM i.e. predose & 12 hours) on each day.
- Estimates of within-subject variability for FeNO will also be provided, where CVw(%) = SQRT(exp(MSE) − 1)×100 and MSE is the residual mean squared error from the model. CVw represents a pooled measure of within-subject variability across the regimens FF/VI 100/25mcg, Placebo and timepoints.

#### **Endpoint**

Change from baseline of FEV1 during treatment with FF/VI.

#### **Secondary Statistical Analyses**

#### **Model Specification**

Endpoints will be statistically analysed using a mixed models repeated measures (MMRM) model.

Terms fitted in the MMRM model will include:

Fixed effect terms: Period, Treatment, Day, Time, Period-level baseline\*Day\*Time interaction term, Treatment\*Day\*Time interaction term, Period-level baseline and Subject-level baseline.

• Repeated: Day\*Time interaction term.

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics will be performed for mentioned Statistical Analyses as required.

#### **Model Results Presentation**

- Point estimates and their associated 95% confidence intervals will be constructed for the difference [FF/VI 100/25mcg] [Placebo] at each timepoint (AM/PM i.e. predose & 12 hours) on each day.
- Estimates of within-subject variability for FEV1 will also be provided, where  $CVw(\%) = SQRT(exp(MSE) 1) \times 100$  and MSE is the residual mean squared error from the model. CVw represents a pooled measure of within-subject variability across the regimens FF/VI 100/25mcg, Placebo and timepoints.

## 9. OTHER STATISTICAL ANALYSES

# 9.1. Overview of Planned Biomarker Analyses

Blood Eosinophil and Serum Periostin levels will be listed and summarised if data is available. The biomarker displays will be based on the "All Subjects" population.

#### 9.1.1. Overview of Planned Analyses

Table 5 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 5 Overview of Planned Biomarker Analyses

| Endpoint | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| • | Summary | | Individual | | Summary | | Individual | |
| | T | F | F | L | T | F | F | L |
| Biomarker | | | | | | | | |
| Biomarker Parameters | Y | | Y | Y | Y | | | |

#### **NOTES:**

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.

| Endpoint | | Ab | solute | ; | Change from Baseline | | | seline |
|---|---|---|---|---|---|---|---|---|
| • | Summary | | Individual | | Summary | | Individual | |
| | T | F | F | L | T | F | F | L |

• Individual = Represents FL related to any displays of individual subject observed raw data.

## 9.2. Overview of Safety Analyses

#### 9.2.1. Overview of Planned Adverse Events Analyses

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 6 Overview of Planned Adverse Event Analyses

| Endpoint | Absolute | | |
|---|---|---|---|
| | Sum | mary | Individual |
| | T | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and PT | Y | | Y |
| Drug-Related AEs by SOC and PT | Y | | |
| Subject Numbers for Individual AEs | | | Y |
| Relationship Between AE SOCs, PT and Verbatim Text | | | Y |
| Serious AEs by SOC and PT | | | Y |
| AEs Leading to Withdrawal from Study / Permanent<br>Discontinuation of Study Treatment by SOC and PT | Y | | Y |

#### **NOTES:**

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 9.2.2. Overview of Planned Clinical Laboratory Analyses

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

 Table 7
 Overview of Planned Clinical Laboratory Analyses

| | Sum | mary | Individual |
|----------------|-----|------|------------|
| | T | F | L |
| Lab Parameters | | | Y |

#### **NOTES:**

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 9.2.3. Overview of Planned Other Safety Analyses

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

 Table 8
 Overview of Planned Other Safety Analyses

| | Sumn | nary | Individual |
|----------------------|------|------|------------|
| | T | F | L |
| Vital Signs by Visit | | | Y |

#### **NOTES:**

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 10. REFERENCES

GlaxoSmithKline Document Number 2015N241692\_00 (Original – 12-JAN-2016): A randomised, placebo-controlled, double-blind, two period crossover study to characterise the exhaled nitric oxide time profile as a biomarker of airway inflammation in adult asthma patients following repeat administration of inhaled Fluticasone Furoate (FF)/ Vilanterol (VI) 100/25 mcg.

# 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | RAP Section 4 : Analysis Populations |
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| | : General Considerations for Data Analyses & Data Handling |
| Conventions | |
| Section 11.2 | Appendix 2: Data Management |
| Section 11.3 | Appendix 3: Time and Events |
| Section 11.4 | Appendix 4 Treatment States & Phases |
| Section 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population |
| Section 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 11.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP Ap | pendices |
| Section 11.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 11.10 | Appendix 10: List of Data Displays |
| Section 11.11 | Appendix 11: Example Mock Shells for Data Displays |

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

As detailed in Section 4.1, Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan and a listing and summary of important Protocol Deviations will be provided. A separate listing and summary of inclusion/exclusion criteria deviations will also be produced based on the eligibility eCRF page.

A Per Protocol Population is not being defined for this study. However additional exploratory sensitivity summaries may be considered, if there are protocol deviations that may affect the primary PD endpoint analysis will be confirmed prior to unblinding. Any additional sensitivity summaries will be documented in the CSR

# 11.2. Appendix 2: Data Management

| Data Type | Source | Format | Planned Date of | Responsibility |
|---|---|---|---|---|
| | | of Data | Final File <sup>1</sup> | |
| <b>Study Population</b> | Database | IDSL | DBF | CPSSO |
| Safety | Database | IDSL | DBF | CPSSO |
| Pharmacodynamic | Database | IDSL | DBF | CPSSO |
| Biomarker | Database | IDSL | DBF | CPSSO |

<sup>1.</sup> Provided source data is clean

# 11.3. Appendix 3: Time & Events

| | Screening (up to | | Study | Day (each tr | reatment per | riod) | | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | 42 days prior to<br>Day 1) | Day -7 (start<br>of run-in) <sup>1</sup> | Day 1 | Days<br>2-13 | Days<br>14-19 | Day<br>21 | Day 35 | (Days 35-<br>42) <sup>12</sup> | |
| Out-patient visit to the unit | X | X | X | | | X | X | X | <sup>1</sup> Day -7 is the start of<br>the one week run-in<br>period and therefore<br>this visit and the<br>assessments on this day<br>only apply to Treatment<br>Period 1 |
| Admission to the unit | | | | | X | | | | |
| Informed consent | X | | | | | | | | |
| Inhaler, PEF meter and FeNO device practice | X | | | | | | | | |
| Inclusion and exclusion criteria/eligibility review | X | X | X | | | | | | |
| Demography | X | | | | | | | | |
| Full physical exam including height and weight | X | | | | | | | | |
| Medical history (includes<br>substance usage [and<br>family history of<br>premature CV disease]) | X | | | | | | | | Substances: [Drugs,<br>Alcohol, tobacco and<br>caffeine] |
| Past and current medical conditions [including cardiovascular medical history] | X | | | | | | | | |

| | Screening (up to | | Study I | Day (each t | reatment per | iod) | | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | 42 days prior to<br>Day 1) | Day -7 (start of run-in) <sup>1</sup> | Day 1 | Days<br>2-13 | Days<br>14-19 | Day<br>21 | Day 35 | (Days 35-<br>42) <sup>12</sup> | |
| Urine pregnancy test (WCBP) | X | | $X^2$ | | | X | | X | <sup>2</sup> Collected pre-dose |
| Vital signs | X | | | | | | | | |
| Set up PEF and FeNO monitoring | | X | | | | | | | |
| Study Treatment | | | Х | 23 | X <sup>4</sup> | | | | <sup>3</sup> Dosing every<br>morning; dosing in the<br>unit on Days 1 and 14<br>and at home on Days 2-<br>13<br><sup>4</sup> Dosing on the<br>morning of Day 14<br>only |
| Exploratory biomarker sampling <sup>5</sup> | | X | | | X | X | X | | <sup>5</sup> These measurements<br>are taken at baseline<br>(Day -7), at the end of<br>treatment (Day 15), on<br>Day 21 and on Day 35. |
| FEV <sub>1</sub> readings <sup>6</sup> | X | | X <sup>7</sup> | | X8 | X <sup>9</sup> | | | <sup>6</sup> Measured in the unit<br>only<br><sup>7</sup> Taken pre-dose<br><sup>8</sup> Collected AM (pre-<br>dose on Day 14) and<br>PM<br><sup>9</sup> Collected AM only |
| FeNO assessment <sup>10</sup> | X | <b>←====</b> | | | | | <del>)</del> | | 10 Start of collection 7<br>days before Day 1 (Day<br>-7), then collected<br>every day AM and PM<br>through to Day 35 of<br>each treatment period. |

| | Screening (up to | | Study 1 | Day (each t | reatment per | iod) | | Follow-up | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | 42 days prior to<br>Day 1) | Day -7 (start<br>of run-in) <sup>1</sup> | Day 1 | Days<br>2-13 | Days<br>14-19 | Day<br>21 | Day 35 | (Days 35-<br>42) <sup>12</sup> | |
| PEF <sup>11</sup> | | <b>←====</b> | | | | | | ====> | 11 Collected AM and PM every day from Day -7 through to Day 35 for Treatment Period 1, and from Day 1 through to follow up for Treatment Period 2. |
| AE/SAE review | | ←===== | | | | | | <del>-</del> | |
| Concomitant medication review | | <b>←</b> | | | | | | → | 12 Follow up visit only after Treatment period 2. The follow-up visit can be combined with the Day 35 visit for Treatment Period 2. |
| Issue of diary card | X | | | | X <sup>13</sup> | | | | 13 Second diary card<br>given out on Day 21 of<br>Treatment Period 1, to<br>capture data for<br>Treatment Period 2 |

# 11.4. Appendix 4: Treatment States and Phases

## 11.4.1. Treatment States for AE Data

| Treatment<br>State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date [+ Lag Time] |
| Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| Onset Time<br>Since 1 <sup>st</sup> Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing]. |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

#### 11.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| R | andAll NG | Data Displays for Reporting | |
| Code | <b>Description Description</b> | | Order [1] |
| A | Placebo | Placebo | 1 |
| В | FF/VI 100/25 mcg | FF/VI 100/25 mcg | 2 |

#### **NOTES:**

1. Order represents treatments being presented in TFL, as appropriate.

#### 11.5.2. Baseline Definition & Derivations

#### 11.5.2.1. Baseline Definitions

For all endpoints (expect as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

| Parameter | Study Assess | ments Consi | Baseline Used in Data | |
|---|---|---|---|---|
| rarameter | Screening | Day -7 | Display | |
| PD | | | | |
| FeNO | X | X | X | Day 1 (Pre-dose) |
| FEV1 | X | | X | Day 1 (Pre-dose) |
| PEF | | X | X | Day 1 (Pre-dose) |
| Biomarker | | | X | Day 1 (Pre-dose) |

• Note: Baseline definitions are applicable to each period

For FeNO, FEV1 analyses:

- Subject level baseline is defined as the mean of baseline across periods for each subject.
- Period level baseline is defined as the difference between the baseline and subject level baseline for each period and each subject.

#### 11.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 11.5.3. Reporting Process & Standards

| <b>Reporting Process</b> | Reporting Process |
|---|---|
| Software | |
| • The currently s | upported versions of SAS software will be used. |
| Reporting Area | Reporting Area |
| HARP Server | : UK1SALX00175-HARP PROD-UK |
| HARP Area | : \ARPROD\ GW685698+GW642444\mid201499\Final |
| QC Spreadsheet | : \ARWORK\ GW685698+GW642444\mid201499\Final\Documents |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards | |
| Generation of RTF Files | |
| • RTF files will b | be generated for summary displays. |

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| | $\mathcal{E}$ |
|---|---|
| <b>Descriptive Summ</b> | ary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Phar | macodynamic Parameters |
| Descriptive Summa | ry N, n, geometric mean, 95% CI of geometric mean, standard |
| Statistics (Log | deviation (SD) of logged data and [between and or within] |
| Transformed) | geometric coefficient of variation (CVb/w (%)) will be reported. |
| | [1] CVb (%) = $\sqrt{\exp(SD2) - 1} * 100$ |
| | (SD = SD of log transformed data) |
| | [2] $CVw$ (%) = $\sqrt{(exp(MSE) - 1) * 100}$ |
| | (MSE = mean square error from mixed effect model of |
| | loge-transformed data). |
| Parameters Not Bei | ng FEV1 |
| Log Transformed | |
| Graphical Displays | |
| • Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 11.6. Appendix 6: Derived and Transformed Data

#### 11.6.1. General

## **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.

#### **Study Day**

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing
- $\rightarrow$  Study Day = Missing
- Ref Date < Treatment start Date → Study Day = Ref Date Treatment start Date
- Ref Data ≥ Treatment start Date → Study Day = Ref Date (Treatment start Date) + 1

#### 11.6.2. Study Population

## **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - o Any subject with a missing day will have this imputed as day '15'.
  - o Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### **Extent of Exposure**

• Number of days of exposure to study drug will be calculated based on the formula:

#### **Duration of Exposure in Days = (Treatment Stop Date – Treatment Start Date) + 1**

- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

**Cumulative Dose = Sum of (Number of Days x Total Daily Dose)** 

#### 11.6.3. Pharmacodynamic

#### **FeNO**

#### Period level baseline

- The Period-Specific Baseline value is the pre-dose assessment collected on day 1 of each treatment period
- Period level baseline is defined as the difference between the baseline and subject level baseline for each period and each subject.

#### Subject level baseline

• Subject level baseline is defined as the mean of baseline across periods for each subject.

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - o Example 1: 2 Significant Digits = < x becomes x 0.01
  - Example 2: 1 Significant Digit = x + 0.1
  - o Example 3: 0 Significant Digits = '< x' becomes x 1

# 11.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

## 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as subject is one who has completed both treatment periods, all assessments up to Day 35 of both treatment periods, and all of the follow-up assessments. The end of the study is defined as the last subject's last visit.</li> <li>Withdrawn subjects were not replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 11.7.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |

# 11.7.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events | <ul> <li>The recorded partial date will be displayed in listings.</li> <li>Any partial dates for adverse events will be raised to data management If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.7.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 11.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### 11.8.1. Statistical Analysis Assumptions

| <b>Endpoint(s)</b> | • | Loge (FeNO) and FEV1 |
|--------------------|---|----------------------|
| Analysis | • | MMRM |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

# 11.9. Appendix 9 – Abbreviations & Trade Marks

## 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| GUI | Guidance |
| MMRM | Mixed Model Repeated Measures |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

## 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |

Trademarks not owned by the GlaxoSmithKline Group of Companies

# 11.10. Appendix 10: List of Data Displays

## 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.10 | - |
| Pharmacodynamic | 2.1 to 2.8 | 2.1 to 2.6 |
| Safety | 3.1 to 3.3 | |
| Biomarker | 4.1 to 4.2 | 4.1 |
| Section | List | tings |
| ICH Listings | 1 to | 18 |
| Other Listings | 19 t | o 25 |

## 11.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|---------------------------|--------|---------|---------|
| Study Population | N/A | POP_Tn | POP_Ln |
| Pharmacodynamic/Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Safety | N/A | SAFE Tn | SAFE Ln |

#### **NOTES:**

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 11.10.3. Deliverable [Priority]

| <b>Delivery Priority</b> | Description |
|--------------------------|-------------------------------------|
| Headline [1] | Headline Results |
| SAC [2] | Final Statistical Analysis Complete |

# 11.10.4. Study Population Tables

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subje | ct Disposition | | | | |
| 1.1. | All Subjects | ES1A | Summary of Subject Disposition for the Subject Conclusion Record | | Headline [1]<br>SAC [2] |
| 1.2. | Screened<br>Subjects | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC [2] |
| 1.3. | Screened<br>Subjects | NS1 | Summary of Number of Subjects by Country and Site ID | | SAC [2] |
| Proto | col Deviation | | | | |
| 1.4. | All Subjects | DV1 | Summary of Important Protocol Deviations | | SAC [2] |
| Popul | ation Analysed | | | | |
| 1.5. | Screened<br>Subjects | SP1 | Summary of Study Populations | | SAC [2] |
| Demo | graphics | | | | |
| 1.6. | All Subjects | DM3 | Summary of Demographic characteristics | Include BMI | Headline [1]<br>SAC [2] |
| 1.7. | PD | DM3 | Summary of Demographic characteristics | Include BMI.<br>Conditional Display | SAC [2] |
| 1.8. | All Subjects | DM11 | Summary of Age Ranges | Include only Adult (18-64) and (65-84) years category | SAC [2] |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.9. | All Subjects | DM5 | Summary of Race and Racial Combinations | | SAC [2] |
| Exposure | | | | | |
| 1.10. | All Subjects | EX1 | Summary of Exposure Data | | SAC [2] |

# 11.10.5. Pharmacodynamic Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| Pharm | acodynamic Pa | rameters | | | |
| 2.1. | PD | LB1 | Summary of Exhaled Nitric Oxide Data | Parameter with units, both untransformed and transformed | Headline [1]<br>SAC [2] |
| 2.2. | PD | LB1 | Summary of Change from Baseline Exhaled Nitric Oxide Data | Parameter with units for untransformed data | SAC [2] |
| 2.3. | PD | LB1 | Summary of Ratio from Baseline Exhaled Nitric Oxide Data | Parameter with units for transformed data | Headline [1]<br>SAC [2] |
| 2.4. | PD | PD_T1 | Summary of Repeated Measures Statistical Analysis of Ratio from Baseline Exhaled Nitric Oxide Data after cessation of repeat dose of treatment | | Headline [1]<br>SAC [2] |
| 2.5. | PD | PD_T1 | Summary of Repeated Measures Statistical Analysis of Ratio from Baseline Exhaled Nitric Oxide Data | | SAC [2] |
| 2.6. | PD | LB1 | Summary of Spirometry data | | SAC [2] |
| 2.7. | PD | LB1 | Summary of Change from Baseline in Spirometry data | | SAC [2] |
| 2.8. | PD | PD_T1 | Summary of Repeated Measures Statistical Analysis of Change from Baseline FEV1 Data | | SAC [2] |

# 11.10.6. Pharmacodynamic Figures

| Phari | nacodynamic: I | Figures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Phari | nacodynamic P | arameters | | | |
| 2.1. | PD | PD_F1 | Plot of Individual Subject of Exhaled Nitric Oxide<br>Time-Profile after cessation of repeat dose<br>treatment | | SAC [2] |
| 2.2. | PD | PD_F2 | Plot of Adjusted Geometric Mean Exhaled Nitric<br>Oxide Ratio from Baseline Time-Profile by<br>Treatment | With confidence intervals taken from repeated measures analysis. Plot to present Day & AM/PM on x-axis and change from baseline ratio on y-axis. One line for each treatment. | Headline [1]<br>SAC [2] |
| 2.3. | PD | PD_F2 | Plot of Exhaled Nitric Oxide Ratio from Baseline<br>Treatment Ratios Against Time | With confidence interval taken from repeated measures analyses. Similar to Figure 2.02 but present treatment ratio instead of adjusted mean. Include horizontal line through 1. | SAC [2] |
| 2.4. | PD | PD_F1 | Plot of Individual Subject of FEV1 Time-Profile | | SAC [2] |
| 2.5. | PD | PD_F2 | Plot of Adjusted Mean FEV1 Change from Baseline Time-Profile by Treatment | With confidence interval taken from repeated measures analysis. Present as for FeNO except present for change from baseline instead of change from baseline ratio. | SAC [2] |
| 2.6. | PD | PD_F2 | Plot of FEV1 Change from Baseline Treatment<br>Differences Against Time | With confidence intervals taken from repeated measures analysis. Present as for FeNO except present for change from baseline instead of change from baseline ratio. | SAC [2] |

# 11.10.7. Safety Tables

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| Adver | se Events | | | | |
| 3.1. | All Subjects | AE1CP | Summary of Adverse Events by System Organ Class and Preferred Term | | Headline [1]<br>SAC [2] |
| 3.2. | All Subjects | AE1CP | Summary of All Drug-Related Adverse Events by<br>System Organ Class and Preferred Term | | SAC [2] |
| 3.3. | All Subjects | AE1CP | Summary of AEs Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | | SAC [2] |

# 11.10.8. Biomarker Tables

| Bioma | Biomarker Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| Bioma | Biomarker parameter | | | | |
| 4.1. | All Subjects | LB1 | Summary of Biomarker Data | | SAC [2] |
| 4.2. | All Subjects | LB1 | Summary of Change from Baseline Biomarker Data | | SAC [2] |

# 11.10.9. Biomarker Figures

| Biomarker: Figure | | | | | |
|---|---|---|---|---|---|
| No. | Population IDSL / Example Title Shell | | Programming Notes | Deliverable<br>[Priority] | |
| Biomark | ker Parameter | | | | |
| 4.1 | PD | PD_F3 | Plot of Histogram of Biomarker Data by<br>Treatment | | SAC [2] |

# 11.10.10. ICH Listings

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Subjec | ct Disposition | | | | |
| 1. | Screened<br>Subjects | ES7 | Listing of Reasons for Screening Failure | | SAC [2] |
| 2. | All Subjects | ES3 | Listing of Reasons for Withdrawal | | SAC [2] |
| 3. | All Subjects | BL2 | Listing of Subjects for Whom the Treatment Blind was Broken During the Study | | SAC [2] |
| 4. | All Subjects | TA2 | Listing of Randomised and Actual Treatments | | SAC [2] |
| Protoc | col Deviations | | | | |
| 5. | All Subjects | DV2A | Listing of all Protocol Deviations | | SAC [2] |
| 6. | All Subjects | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [2] |

| ICH: | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Subject | ct Disposition | | | | |
| 7. | Screened<br>Subjects | SP3A | Listing of Subjects Excluded from Any Population | | SAC [2] |
| Demo | graphics | | | | |
| 8. | All Subjects | DM4 | Listing of Demographic Characteristics | | SAC [2] |
| 9. | All Subjects | DM10 | Listing of Race | | SAC [2] |
| Prior | and Concomita | ant Medication | | | |
| 10. | All Subjects | MH2 | Listing of Medical Conditions | isting of Medical Conditions | |
| 11. | All Subjects | CP_CM4 | Listing of Concomitant Medications by Generic Terms | SAC [2] | |
| Expos | ure | | | | |
| 12. | All Subjects | EX4 | Listing of Exposure Data | | SAC [2] |
| AE | | | | | |
| 13. | All Subjects | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC [2] |
| 14. | All Subjects | AE9CP | Listing of All Adverse Events | | SAC [2] |
| 15. | All Subjects | AE9CP | Listing of Serious Adverse Events | | SAC [2] |
| 16. | All Subjects | AE9CP | Listing of AEs Leading to Withdrawal from Study | | SAC [2] |
| Vitals | /LAB | | | | |
| 17. | All Subjects | VS5 | Listing of Vital Signs | | SAC [2] |
| 18. | All Subjects | CP_LB6 | Listing of Laboratory Data for Subjects | | SAC [2] |

# 11.10.11. Non-ICH Listings

| Non-I | CH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| AE | | | | | |
| 19. | All Subjects | AE2 | Listing of Relationship between System Organ Class and Verbatim Text | | SAC [2] |
| Pharm | nacodynamic/F | Biomarker | | | |
| 20. | PD | EG4 | Listing of Exhaled Nitric Oxide Data | | SAC [2] |
| 21. | PD | EG4 | Listing of Spirometry Data | | SAC [2] |
| 22. | PD | EG4 | Listing of Biomarker Data | | SAC [2] |
| 23. | PD | | Raw SAS Output from Repeated Measures Statistical Analysis of Change from Baseline RatioExhaled Nitric Oxide Data after cessation of repeat dose treatment | | SAC [2] |
| 24. | PD | | Raw SAS Output from Repeated Measures Statistical Analysis of Change from Baseline RatioExhaled Nitric Oxide Data | | SAC [2] |
| 25. | PD | | Raw SAS Output from Repeated Measures Statistical Analysis of Change from Baseline FEV1 | | SAC [2] |

#### **CONFIDENTIAL**

201499

# 11.11. Appendix 11: Example Mock Shells for Data Displays

Example : PD\_T1 Page 1 of 2

Protocol : 201499 Population : PD

Table 2.3

Summary of Repeated Measures Statistical Analysis of Ratio from Baseline Exhaled Nitric Oxide Data after cessation of repeat dose of treatment

| Parameter | Visit | Planned<br>Timepoint | Comparison | Adjusted Geometric<br>Mean | | Geometric | | Ratio (Test/Ref) | 95% Confidence Interval for Ratio | %CVw |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | n | Test | n | Ref | (Test/Itel) | | |
| FeNO | | | Test vs Ref | X | XX.XX | X | XX.XX | X.XXXX | (x.xxxx, x.xxxx) | XX.X |

Example : PD\_F1 

Protocol : 201499 Population : PD

Figure 2.1.

Plot of Individual Subject of Exhaled Nitric Oxide Time-Profile after cessation of repeat dose treatment



Plot to present Day & AM/PM on x-axis and PD endpoints on y-axis. One line for each treatment.

Example : PD\_F2 

Protocol : 201499 Population : PD

Figure 2.2

Plot of Adjusted Geometric Mean Exhaled Nitric Oxide Ratio from Baseline Time-Profile by Treatment



Plot to present Day & AM/PM on x-axis but change from baseline ratio on y-axis. One line for each treatment.

Example : PD\_F3 

Protocol : 201499 Population : PD

Figure 4.1
Plot of Histogram of Biomarker Data by Treatment

